CLINICAL TRIAL: NCT04562415
Title: The Effect Of Sham Controlled Continuous Theta Burst Stimulation And Low Frequency Repetitive Transcranial Magnetic Stimulation On Upper Extremity Spasticity And Functional Recovery In Patients With Ischemic Stroke
Brief Title: The Effect Of Transcranial Magnetic Stimulation In Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Clinical Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2020-09-19; First posted 2020-09-24 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: Stroke; Repetitive Transcranial Magnetic Stimulation; Continuous Theta Burst Stimulation; Functional Recovery; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active rTMS group (Active Comparator): chronic ischemic stroke patients receiving active low frequency repetitive transcranial magnetic stimulation therapy and physical therapy
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation Therapy
- Active cTBS group (Active Comparator): chronic ischemic stroke patients receiving active continuous theta burst stimulation therapy and physical therapy
  Interventions: Device: Active Continuous Theta Burst Stimulation Therapy
- Sham cTBS group (Sham Comparator): chronic ischemic stroke patients receiving sham continuous theta burst stimulation therapy and physical therapy
  Interventions: Device: Sham Continuous Theta Burst Stimulation Therapy

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation Therapy — 10 sessions of intact hemispheric upper extremity motor area (M1) were targeted and inhibitor rTMS was applied with a frequency of 1 Hz consisting of 1200 pulses for 20 minutes. In addition, within 30 minutes after TMS sessions, all patients underwent 10 sessions of joint range of motion, stretching, strengthening, balance and coordination exercises, hand rehabilitation and daily living activities.
  Other Names: Rehabilitation Program
  Arms: Active rTMS group
Device: Active Continuous Theta Burst Stimulation Therapy — 10 sessions of intact hemispheric upper extremity motor area (M1) were targeted and cTBS was administered for a total of 600 pulses consisting of 3 burst stimulations of 50 Hz repeated every 200 milliseconds for 40 seconds. In addition, within 30 minutes after TMS sessions, all patients underwent 10 sessions of joint range of motion, stretching, strengthening, balance and coordination exercises, hand rehabilitation and daily living activities.
  Other Names: Rehabilitation Program
  Arms: Active cTBS group
Device: Sham Continuous Theta Burst Stimulation Therapy — 10 sessions of intact hemispheric upper extremity motor area (M1) were targeted and sham cTBS was administered for a total of 600 pulses consisting of 3 burst stimulations of 50 Hz repeated every 200 milliseconds for 40 seconds. In addition, within 30 minutes after TMS sessions, all patients underwent 10 sessions of joint range of motion, stretching, strengthening, balance and coordination exercises, hand rehabilitation and daily living activities.
  Other Names: Rehabilitation Program
  Arms: Sham cTBS group

SUMMARY:
This study is aimed to investigate the effect of continuous theta burst stimulation (cTBS) and low frequency repetitive transcranial magnetic stimulation (rTMS) on upper extremity spasticity and functional recovery in patients with chronic ischemic stroke.

DETAILED DESCRIPTION:
A sham-controlled double-blind randomized study was undertaken. 20 patients with chronic stroke were randomized into active rTMS group (n=7), active cTBS group (n=7) and sham cTBS group (n=6). In the active rTMS group, 10 sessions of intact hemispheric upper extremity motor area (M1) were targeted and inhibitor rTMS was applied with a frequency of 1 Hz consisting of 1200 pulses for 20 minutes. In the active cTBS group, 10 sessions of intact hemispheric upper extremity motor area (M1) were targeted and cTBS was administered for a total of 600 pulses consisting of 3 burst stimulations of 50 Hz repeated every 200 milliseconds for 40 seconds. Sham cTBS was applied in the same protocol but using sham coil. Within 30 minutes after TMS sessions, all patients underwent 10 sessions of joint range of motion, stretching, strengthening, balance and coordination exercises, hand rehabilitation and daily living activities under the guidance of a physiotherapist, regardless of which group they were in. Upper Extremity Fugl-Meyer Motor Function Scale, Modified Ashworth Scale (MAS), Functional Independence Measure (FIM), Motor Activity Log-28 (MAL-28) and Brunnstrom upper extremity and hand motor recovery stage were assessed at pre-treatment, post-treatment and follow up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke with a disease interval of 6 months to 2 years
* aged between 18-80 years
* Mini mental test score ≥ 24
* upper limb Brunnstrom recovery stage 3 to 5
* upper extremity (elbow, wrist and finger) spasticity level Modified Ashworth Scale (MAS) 1+ to 3

Exclusion Criteria:

* hemorrhagic stroke
* history of epilepsy
* a cardiac pacemaker
* pregnancy
* history of previous stroke or ischemic attack
* neurological diseases other than stroke
* metallic implant in brain or scalp (including cochlear implant)
* previous brain surgery
* orthopedic disease that prevents upper extremity movements
* poor general health (due to heart failure, chronic obstructive pulmonary disease, severe infection, etc.)
* diagnosis of malignancy
* injections of botulinum toxin in the last 6 months for the affected upper extremity
* drug or dosage changes of anti-spasticity medications in the last 1 month period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Fugl-Meyer Motor Function Scale | up to 6 weeks
  Scale measures level of upper extremity motor functions (min-max: 18-126 points). Higher values represent a better outcome.
Modified Ashworth Scale | up to 6 weeks
  Scale measures muscle tone (spasticity) (min-max:0-4). Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Functional Independence Measure | up to 6 weeks
  Scale measures level of independence on activities of daily life (min-max: 18-126 points). Self-care part of the motor subscale was used in this study (min-max:6-42 points). Higher values represent a better outcome.
Motor Activity Log-28 | up to 6 weeks
  Scale measures frequency of use and functionality level of the affected upper limb during daily activities (min-max: 0-5 points). Higher values represent a better outcome.
Brunnstrom Motor Recovery Scale | up to 6 weeks
  Scale measures upper extremity and hand motor recovery stages (min-max: 1-6). Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Yılmaz, Professor,MD, Study Director — Gaziler PMR, Training and Research Hospital, Department of PMR; Ömer Kuzu, MD, Principal Investigator — Gaziler PMR, Training and Research Hospital, Department of PMR
Locations (1):
- Gaziler PMR, Training and Research Hospital, Department of PMR, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No